CLINICAL TRIAL: NCT01888939
Title: Effects of Interrupting Sedentary Behavior on Metabolic and Cognitive Outcomes in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130169; 13-CH-0169
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01-29

CONDITIONS: Healthy Volunteer
Keywords: Executive Function; Child; Obesity; Exercise; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance

INTERVENTIONS:
Other: Walking on a Treadmill
Other: Sedendary Activities Only

SUMMARY:
Background:

- Some studies in adults have found that insulin and glucose blood levels are lower when a long period of sitting is broken up with walking, compared to sitting without breaks. This means that the body can better process sugars when there are walking breaks during the day. Researchers want to know if this is also true for children. Some studies have found that children s attention and memory might be better after exercise. Researchers want to know if short walking breaks have the same effects.

Objectives:

- To understand if breaking up sitting with walking helps children s bodies better use sugars and improves children s concentration.

Eligibility:

- Healthy children ages 7 to 11.

Design:

* Participants will be screened with a physical exam, medical history, exercise test, picture vocabulary test, and medical tests including blood tests and X-rays.
* Participants will return for two 7-hour visits. In the month before the visits, they will wear a physical activity monitor for one week so researchers know how active they are. Once they will take the sitting only test and once the sitting breaks test.
* During the sitting only test, participants will sit for 3 hours.
* During the sitting breaks test, they will sit for 3 hours with 3-minute walking breaks every 30 minutes.
* Both days, they will drink sugar water. Then the participants will have blood drawn from a needle that is kept in place, and they will wear a heart monitor. They will take attention and working memory tests on a computer and answer questions about how they feel. They will eat a meal at the end of the test day.

DETAILED DESCRIPTION:
Prevention of pediatric obesity and its complications are U.S. public health priorities. Promoting physical activity has been proposed as an intervention strategy. Apart from reducing excessive weight, physical activity improves cardiovascular fitness, insulin sensitivity, and academic performance. However, emerging evidence in adults suggests that increased physical activity may not entirely counteract the negative health effects of a sedentary lifestyle.

Sedentary behavior is defined as a set of low-intensity activities involving limited body movement (e.g.: TV viewing, prolonged sitting). TV viewing is associated with lower cognitive functioning and depressive symptoms. Some studies found higher levels of childhood sedentary behavior predicted higher body mass index (BMI) and cholesterol in adulthood, suggesting that negative health consequences may begin early. Dunstan et al. conducted the first lab-based study in adults investigating interrupting prolonged sedentary behavior with physical activity breaks. The authors found that for overweight adults, adding 2-minute moderate-intensity walking breaks every 20 minutes reduced postprandial insulin and glucose responses by 23.0% and 29.6%, respectively. Thus, interrupting sedentary behavior may be an intervention strategy to reduce health risks.

In children, cross-sectional observational studies indicate that sedentary behavior patterns characterized by short bouts of activity are not associated with increased cardiometabolic risk. However to date, no in-lab studies have manipulated sedentary behavior in children. Therefore, we propose to conduct a randomized crossover pilot feasibility study to assess whether interrupting sedentary behavior influences metabolic and executive function, attention, mood, anxiety, and dietary intake. Children, ages 7-11 years, will complete two conditions in random order: 3 hours of prolonged sitting and 3 hours of sitting interrupted with 3 minutes of moderate-intensity walking every 30 minutes. The specific aim of this project is to investigate whether interrupting sedentary behavior improves metabolic parameters and changes executive function, attention, mood, anxiety, and dietary intake. The primary hypothesis is that postprandial insulin incremental area under the curve (iAUC) will be lower in the interrupted sitting vs. the prolonged sitting condition. The exploratory secondary hypotheses are that glucose iAUC, executive function, attention, mood, anxiety, and dietary intake will differ between the two conditions.

This project will investigate if interrupting sedentary time affects potential negative health consequences of sedentary behavior in children. If interrupting sedentary time in short bouts has beneficial effects among children, interventions examining the frequency, duration, and intensity of such interruptions could be developed. Thus, these results have the potential to provide insight into novel behavioral intervention targets in youth.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will qualify for the study if they meet the following criteria:

1. Good general health.
2. Age greater than or equal to 7 and <11.99 years.
3. Fasting plasma glucose < 100 mg/dL
4. a) Phase 1: Body mass index (BMI) between the 5th and 85th percentiles, as determined by the CDC age- and sex- specific growth charts.

   b) Phase 2: BMI above the 85th percentile, as determined by the CDC age- and sex- specific growth charts.

EXCLUSION CRITERIA:

1. Significant cardiac or pulmonary disease likely to or resulting in hypoxia or decreased perfusion.
2. Evidence of impaired glucose tolerance or type 2 diabetes, including fasting plasma glucose greater than or equal to 100 mg/dL.
3. Presence of other endocrinologic disorders leading to obesity (e.g.: Cushing Syndrome).
4. Participants who have, or whose parent/guardians have, current substance abuse or a psychiatric disorder or other condition that, in the opinion of the investigators, would impede competence, compliance, or prevent the completion of the study.
5. Participants who have, or are currently receiving, anti-psychotic drugs that would affect metabolism, cognitive outcomes, and body habitus.
6. Participants receiving medical treatment other than diet for hypertension or dyslipidemia.
7. Participants with precocious puberty and/or receiving androgen and estrogen therapy.
8. Participants currently taking medications for ADHD, or any disorder or use of medications known to affect body composition or weight.
9. Presence of pre-existing neurocognitive disabilities, or an age-adjusted score below 85 on the Picture Vocabulary Test at the screening visit.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2013-06-26; Primary Completion 2017-03-08 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Lower insulin incremental area under the curve (iAUC) during 3 hours after the OGTT. | 3 hours

SECONDARY OUTCOMES:
Lower postprandial glucose iAUC during 3 hours after the OGTT. | 3 hours
Differences in executive functioning and attention scores. | 3 hours
Differences in positive and negative affect scores. | 3 hours
Differences in anxiety. | 3 hours
Differences in post-test dietary intake. | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z, Wei R, Curtin LR, Roche AF, Johnson CL. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11. 2002 May;(246):1-190. PMID 12043359
- [Background] Jago R, Harrell JS, McMurray RG, Edelstein S, El Ghormli L, Bassin S. Prevalence of abnormal lipid and blood pressure values among an ethnically diverse population of eighth-grade adolescents and screening implications. Pediatrics. 2006 Jun;117(6):2065-73. doi: 10.1542/peds.2005-1716. PMID 16740849
- [Background] Ventura E, Davis J, Byrd-Williams C, Alexander K, McClain A, Lane CJ, Spruijt-Metz D, Weigensberg M, Goran M. Reduction in risk factors for type 2 diabetes mellitus in response to a low-sugar, high-fiber dietary intervention in overweight Latino adolescents. Arch Pediatr Adolesc Med. 2009 Apr;163(4):320-7. doi: 10.1001/archpediatrics.2009.11. PMID 19349560
- [Derived] Belcher BR, Berrigan D, Papachristopoulou A, Brady SM, Bernstein SB, Brychta RJ, Hattenbach JD, Tigner IL Jr, Courville AB, Drinkard BE, Smith KP, Rosing DR, Wolters PL, Chen KY, Yanovski JA. Effects of Interrupting Children's Sedentary Behaviors With Activity on Metabolic Function: A Randomized Trial. J Clin Endocrinol Metab. 2015 Oct;100(10):3735-43. doi: 10.1210/jc.2015-2803. Epub 2015 Aug 27. PMID 26312582